CLINICAL TRIAL: NCT06109792
Title: Patient Satisfaction and Oral Health-related Quality of Life (OHRQL) For Two Pick-up Techniques of the Locator Retentive Caps for Two Implant-supported Mandibular Overdentures: A Crossover Study
Brief Title: Patient Satisfaction and Oral Health-related Quality of Life (OHRQL) For Two Pick-up Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A0108023RP
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Prosthesis User

STUDY DESIGN:
Intervention Model Description: Group I: Ten overdentures with locator retentive caps and blue inserts were picked up by the indirect method.
  Group II: Ten overdentures with locator retentive caps and pink inserts were picked up by the indirect method.
  Group III: Ten overdentures with locator retentive caps and blue inserts were picked up by the direct method.
  Group IV: Ten overdentures with locator retentive caps and pink inserts were picked up by the direct method.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- • Group I (Active Comparator): Ten overdentures with locator retentive caps and blue inserts were picked up by the indirect method.
  Interventions: Procedure: implant supported mandibular overdenture
- • Group II (Active Comparator): Ten overdentures with locator retentive caps and pink inserts were picked up by the indirect method.
  Interventions: Procedure: implant supported mandibular overdenture
- Group III (Active Comparator): Ten overdentures with locator retentive caps and blue inserts were picked up by the direct method.
  Interventions: Procedure: implant supported mandibular overdenture
- Group IV (Active Comparator): Ten overdentures with locator retentive caps and pink inserts were picked up by the direct method.
  Interventions: Procedure: implant supported mandibular overdenture

INTERVENTIONS:
Procedure: implant supported mandibular overdenture — In this crossover study, the patients received overdentures with two successive different pick-up techniques for the locator retentive caps; each technique was evaluated for patient satisfaction with blue and pink retentive inserts.

SUMMARY:
This study aimed to evaluate patient satisfaction and OHRQL using two pick-up methods for locator retained mandibular overdenture

ELIGIBILITY:
Inclusion Criteria:

* 1. All selected patients will have two implants placed in the mandibular interforaminal region.

  2. All selected patients have a healthy mucosa and have no clinical complications.

  3. All patients are cooperative and approve of the proposed treatment protocol

Exclusion Criteria:

* 1. Patients who refuse to participate in the study 2.Patients who need implant placement as a result of previous implant failure

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | One year
  patient satisfaction was recorded using score system on a scale from 0 to 100
oral health related quality of life | one year
  Oral health related quality of life was evaluated by using scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University ,Faculty of dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No